CLINICAL TRIAL: NCT01122836
Title: Dosing Study of Massage for Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01AT004411-02 (NIH)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Chronic Neck Pain
Keywords: Massage; Chronic Neck Pain; Dosing Study
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Massage Dose 1 (Experimental): This arm receives weekly 60-minute massage for 4 weeks after a 4-week period of no treatment.
  Interventions: Other: Massage
- Massage - Dose 2 (Experimental): This arm receives weekly 60-minute massage for 4 weeks.
  Interventions: Other: Massage
- Massage - Dose 3 (Experimental): This arm receives 2 weekly 30-minute massage for 4 weeks.
  Interventions: Other: Massage
- Massage - Dose 4 (Experimental): This arm receives 2 weekly 60-minute massages for 4 weeks.
  Interventions: Other: Massage
- Massage - Dose 5 (Experimental): This arm receives 3 weekly 30-minute massages for 4 weeks.
  Interventions: Other: Massage
- Massage - Dose 6 (Experimental): This arm receives 3 weekly 60-minute massages for 4 weeks.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Therapeutic Massage

SUMMARY:
This study is designed to determine the most effective dose of massage for persons with chronic neck pain. This information is necessary before more definitive studies can be conducted.

DETAILED DESCRIPTION:
This study's long-term objective is to identify effective treatments for with neck pain. Many Americans have found conventional medical treatments ineffective for this common and costly problem and are increasingly trying complementary and alternative treatments, including therapeutic massage. Despite the growing popularity of massage, its effectiveness for treating neck pain remains unclear, largely because of the poor quality of research in this area. A major deficiency of previous studies has been their use of low "doses" of massage that massage therapists consider inadequate. Unfortunately, the numbers of minutes per massage session, sessions per weeks, or weeks of treatment necessary for massage to have beneficial or optimal effects are not known. This study is designed to address these gaps in our knowledge by determining, for persons with chronic neck pain: 1) the optimal combination of number of treatments per week and length of individual treatment session, and 2) the optimal number of weeks of treatment. In this project, 228 persons with chronic non-specific neck pain will be randomized to a wait list control group or 4 weeks of treatment with one of 5 different dosing combinations (2 or 3 30-minute treatments per week or 1, 2, or 3 60-minute treatments per week). At the end of this 4 week primary treatment period, participants initially receiving each of the 5 dosing combinations will be randomized to a secondary treatment period of either no additional treatment or 6 weekly 60-minute massages. The primary outcomes, neck-related dysfunction and pain, will be assessed by blinded telephone interviewers 4, 10, and 26 weeks post-randomization. To better characterize the trajectory of the persistence of treatment effects, these interview data will be supplemented with outcomes data collected by mailed questionnaire at 8, 14, 18 and 39 weeks. Comparisons of outcomes for the 6 groups during the primary treatment period will identify the optimal weekly dose, while comparisons of outcomes during the secondary treatment period will determine if 10 weeks of treatment is superior to 4 weeks. The results of this study will: 1) guide the development of a massage treatment protocol to be used in a full-scale trial evaluating the effectiveness of therapeutic massage for chronic neck pain, 2) serve as a model for future dosing studies of massage and bodywork, and 3) help interpret the adequacy of the dosing of massage used in past studies of massage for neck pain

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with non-specific, uncomplicated neck pain of at least moderate level of pain
* Lives or works within Greater Seattle WA geographic area

Exclusion Criteria:

* Cervical Radiculopathy
* History of cancer (other than nonmelanoma skin cancer)
* Severe disk problems
* Unstable medical conditions
* Previous neck surgery
* Physically unable to get on and off of a massage table
* Has had massage within the last year
* Currently in litigation for neck pain
* Seeking other treatment for neck pain
* Potential contraindications for massage
* Unable to give informed consent

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement in neck related dysfunction | 4 weeks
  Evidence of clinically important improvement according to the Neck Pain Disability Index
Improvement in pain levels | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Sherman, MPH, PhD, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

REFERENCES:
- [Derived] Cook AJ, Wellman RD, Cherkin DC, Kahn JR, Sherman KJ. Randomized clinical trial assessing whether additional massage treatments for chronic neck pain improve 12- and 26-week outcomes. Spine J. 2015 Oct 1;15(10):2206-15. doi: 10.1016/j.spinee.2015.06.049. Epub 2015 Jun 19. PMID 26096474
- [Derived] Sherman KJ, Cook AJ, Kahn JR, Hawkes RJ, Wellman RD, Cherkin DC. Dosing study of massage for chronic neck pain: protocol for the dose response evaluation and analysis of massage [DREAM] trial. BMC Complement Altern Med. 2012 Sep 18;12:158. doi: 10.1186/1472-6882-12-158. PMID 22985134